CLINICAL TRIAL: NCT03230006
Title: Efficacy Evaluation of Transdiagnostic CBT for Comorbid Alcohol Use and Anxiety Disorders
Brief Title: Transdiagnostic CBT for Comorbid Alcohol Use and Anxiety Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Todd Farchione, Research Associate Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AA023676 (NIH)
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Results first posted 2025-02-25 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Alcohol Use Disorder; Anxiety Disorders
MeSH Terms: conditions — Alcoholism; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two conditions: 1) treatment with the UP or 2) treatment with therapist-guided Take Control (TC; a computerized alcohol reduction program). In addition, in a subset of twenty-five participants, functional magnetic resonance scanning (fMRI) will be used to examine the effects of the UP on changes in brain activity in areas important to regulation of emotional and reward processes implicated in excessive alcohol consumption.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unified Protocol (Active Comparator): The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders (UP) consists of 5 core skills modules based on cognitive behavioral treatment elements of proven effectiveness. As noted above, these core skills modules were designed to target (and have been shown to address) negative emotionality and aversive reactivity to emotional experiences when they occur. These modules are preceded by an introductory session that reviews the patient's presenting symptoms and provides a therapeutic rationale, as well as a module on motivational enhancement. A final module consists of relapse prevention. As the treatment proceeds, the domains of thoughts, feelings, and behaviors are each explored in detail, focusing specifically on elucidating dysfunctional emotion regulation strategies that the patient has developed over time within each of these domains, and teaching patients more adaptive emotion regulation skills.
  Interventions: Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders
- Take Control (Placebo Comparator): TC is a psychotherapy platform derived from the National Institute on Alcohol Abuse and Alcoholism's (NIAAA) self-help approach, Rethinking Drinking. In this study, TC, originally designed as a computerized treatment has been modified to be administered by the therapist to control for effects that may be related to patient-therapist interaction (as opposed to elements of the treatment itself).
  Interventions: Behavioral: Take Control

INTERVENTIONS:
Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders — The UP will be conducted in a standardized fashion over 16 sessions, in a minimum of 16- and a maximum of 21-weeks, following the published therapist guide with minor refinements for application in the proposed comorbid population.
  Other Names: UP
  Arms: Unified Protocol
Behavioral: Take Control — TC will be conducted over 12 sessions, in a minimum of 12- and a maximum of 16-weeks. Therapists will review material from TC and offer general advice on implementation of the alcohol reduction skills in daily life.
  Other Names: TC
  Arms: Take Control

SUMMARY:
Almost 18 million US adults have alcohol use disorders (AUD), with one third of these individuals also diagnosed with anxiety disorders (AXD). The coexistence of AUD and AXD imposes a high burden via healthcare costs and lost productivity. To date, existing treatment approaches for addressing AUD/AXD comorbidity have been only modestly effective and there is a lack of adequate research to guide treatment decisions.

The Unified Protocol (UP) is a transdiagnostic, cognitive-behavioral therapy that has shown efficacy in treating emotional disorders. The efficacy of the UP to facilitate abstinence from alcohol consumption in individuals with comorbid AUD/AXD has also been examined, with results from this study indicating a reduction from baseline in drinks consumed per day. However, further evaluation of the UP for managing AUD/AXD is warranted.

In this clinical trial, the investigators will further assess the UP's effectiveness in reducing alcohol consumption in patients with comorbid AUD/AXD. Participants will be randomized to one of two conditions: 1) treatment with the UP or 2) treatment with therapist-guided Take Control (TC; a computerized alcohol reduction program). In addition, in a subset of twenty-five participants, functional magnetic resonance scanning (fMRI) will be used to examine the effects of the UP on changes in brain activity in areas important to regulation of emotional and reward processes implicated in excessive alcohol consumption.

The researchers' primary hypotheses are that the UP group will, compared to the TC group: 1) be superior in acute symptom reduction from pre- to post-treatment, and 2) evidence greater reductions in percent days heavy drinking, percent days of drinking per week, and alcohol craving.

ELIGIBILITY:
1. DSM-5 diagnosis of an alcohol use disorder (AUD)
2. DSM-5 diagnosis of Social Anxiety Disorder (SAD), Panic Disorder/Agoraphobia (PD/A), Generalized Anxiety Disorder (GAD), and/or Obsessive Compulsive Disorder (OCD) as determined by a clinician-administered diagnostic assessment using the Anxiety Disorder Interview Schedule (ADIS) for the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5); and are rated as crossing the threshold for a formal DSM-5 diagnosis by assignment of an ADIS clinical severity rating (CSR) of 4 (definitely disturbing/disabling on the 0-8 CSR scale) or higher on at least the principal diagnosis.
3. Adults 21 years old or older
4. Expressed desire to stop drinking alcohol completely or to reduce alcohol consumption
5. Reported drinking an average of at least 15 standard drinks per week for males, or 8 for females occurring over a 28-consecutive day period during the 90 day-long time window that preceded the screening session
6. Must be willing to discontinue any form of psychotherapy, except Alcoholics Anonymous (AA), that he or she may be receiving for either anxiety or depression prior to screening.

Exclusion Criteria:

1. DSM-5 diagnosis of current major depressive disorder (with the exception of substance-induced depressive disorder) that requires immediate treatment with pharmacologic agents, bipolar disorder, schizophrenia, current bulimia/anorexia, dementia, or other substance dependence, with the exception of nicotine, marijuana, and caffeine dependence.
2. Presence of suicidal ideation or history of suicide attempts
3. Non-English speakers
4. Previously received an adequate trial of cognitive-behavioral therapy (CBT; 8 sessions within the past 5 years)
5. Contraindications to MRI scans
6. History of head injury with >5-minute loss of consciousness
7. Pregnancy Note: Women of childbearing potential (not postmenopausal for at least one year) will be required to provide a negative urine pregnancy test prior to each scan.
8. Implantation of anything containing magnetically sensitive material including metal plates, aneurysm clips, and cardiac pacemakers, stents; history of sheet metal work, claustrophobia
9. Cognitive impairment (MOCA<21).
10. Serious medical illness or instability for which hospitalization may be likely within the next year.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Farchione, PhD, Principal Investigator — Boston Univeristy
Locations (1):
- Boston University, Charles River Campus, Boston, Massachusetts, United States

REFERENCES:
- [Background] Sauer-Zavala S, Boswell JF, Gallagher MW, Bentley KH, Ametaj A, Barlow DH. The role of negative affectivity and negative reactivity to emotions in predicting outcomes in the unified protocol for the transdiagnostic treatment of emotional disorders. Behav Res Ther. 2012 Sep;50(9):551-7. doi: 10.1016/j.brat.2012.05.005. Epub 2012 Jun 9. PMID 22738907
- [Background] Boswell JF, Farchione TJ, Sauer-Zavala S, Murray HW, Fortune MR, Barlow DH. Anxiety sensitivity and interoceptive exposure: a transdiagnostic construct and change strategy. Behav Ther. 2013 Sep;44(3):417-31. doi: 10.1016/j.beth.2013.03.006. Epub 2013 Apr 2. PMID 23768669

RESULTS

PARTICIPANT FLOW:
Groups:
- Unified Protocol: The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders (UP) consists of 5 core skills modules based on cognitive behavioral treatment elements of proven effectiveness. As noted above, these core skills modules were designed to target (and have been shown to address) negative emotionality and aversive reactivity to emotional experiences when they occur. These modules are preceded by an introductory session that reviews the patient's presenting symptoms and provides a therapeutic rationale, as well as a module on motivational enhancement. A final module consists of relapse prevention. As the treatment proceeds, the domains of thoughts, feelings, and behaviors are each explored in detail, focusing specifically on elucidating dysfunctional emotion regulation strategies that the patient has developed over time within each of these domains, and teaching patients more adaptive emotion regulation skills.
  The UP will be conducted in a standardized fashion, over 16 sessions, following the published therapist guide with minor refinements for application in the proposed comorbid population.
- Take Control: TC is a psychotherapy platform derived from the National Institute on Alcohol Abuse and Alcoholism's (NIAAA) self-help approach, Rethinking Drinking. In this study, TC, originally designed as a computerized treatment has been modified to be administered by the therapist to control for effects that may be related to patient-therapist interaction (as opposed to elements of the treatment itself). Specifically, over 12 sessions on a weekly basis, therapists will review material from TC and offer general advice on implementation of the alcohol reduction skills in daily life.
Period: Overall Study
Arm/Group | Unified Protocol | Take Control
Started | 51 | 24
Completed | 38 | 21
Not Completed | 13 | 3

BASELINE CHARACTERISTICS:
Groups:
- Take Control: Take Control (TC) is a psychotherapy platform derived from the National Institute on Alcohol Abuse and Alcoholism's (NIAAA) self-help approach, Rethinking Drinking. In this study, TC, originally designed as a computerized treatment has been modified to be administered by the therapist to control for effects that may be related to patient-therapist interaction (as opposed to elements of the treatment itself). Specifically, on a weekly basis for 12 sessions, therapists will review material from TC and offer general advice on implementation of the alcohol reduction skills in daily life.
- Total: Total of all reporting groups
Arm/Group | Unified Protocol | Take Control | Total
Number analyzed (Participants) | 51 | 24 | 75
Age, Continuous [Mean (Full Range); unit: Years] | 43.71 [24 to 71] | 41.83 [21 to 66] | 43.11 [21 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 15 | 44
  Male | 22 | 9 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 48 | 23 | 71
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 39 | 22 | 61
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 51 | 24 | 75

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Drinks Consumed Per Week
Description: The Timeline Followback (TLFB) was used to estimate participants' daily drinking during the 90-day period preceding the baseline assessment and was subsequently administered at the beginning of each psychotherapy session and during the follow-up sessions.
Time Frame: Change from baseline following 12-sessions (Take Control Arm), up to 16 weeks, or 16-sessions (Unified Protocol Arm), up to 21 weeks, of treatment.
Population: Analyses were carried out using one-way repeated measures ANOVAs. This type of analysis only includes data from participants who completed treatment, and excludes non-completers.
Measure: Mean (Standard Deviation); unit: Standard Drinking Units per Week
Groups:
- Unified Protocol: The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders (UP) consists of 5 core skills modules based on cognitive behavioral treatment elements of proven effectiveness. As noted above, these core skills modules were designed to target (and have been shown to address) negative emotionality and aversive reactivity to emotional experiences when they occur (Boswell et al., 2013; Carl et al., 2014; Sauer-Zavala et al., 2012). These modules are preceded by an introductory session that reviews the patient's presenting symptoms and provides a therapeutic rationale, as well as a module on motivational enhancement. A final module consists of relapse prevention. As the treatment proceeds, the domains of thoughts, feelings, and behaviors are each explored in detail, focusing specifically on elucidating dysfunctional emotion regulation strategies that the patient has developed over time within each of these domains, and teaching patients more adaptive emotion regulation skills.
  The UP will be conducted in a standardized fashion, over 16 sessions, following the published therapist guide with minor refinements for application in the proposed comorbid population.
- Take Control: TC is a psychotherapy platform derived from the National Institute on Alcohol Abuse and Alcoholism's (NIAAA) self-help approach, Rethinking Drinking. In this study, TC, originally designed as a computerized treatment has been modified to be administered by the therapist to control for effects that may be related to patient-therapist interaction (as opposed to elements of the treatment itself). Specifically, on a weekly basis, for 12 sessions, therapists will review material from TC and offer general advice on implementation of the alcohol reduction skills in daily life.
Arm/Group | Unified Protocol | Take Control
Number analyzed (Participants) | 51 | 24
Standard Drinking Units per Week
  Weekly Average Drinks at Baseline | 40.82 (49.07) | 29.62 (20.09)
  Weekly Average Drinks at Post-Treatment: number analyzed (Participants) | 38 | 21
  Weekly Average Drinks at Post-Treatment | 12.12 (10.89) | 23.86 (21.54)
Statistical Analysis 1: Comparison: Unified Protocol vs Take Control; Test type: Superiority; p = 0.002, ANOVA; Partial eta squared = .152 — A two-way mixed ANOVA was conducted to investigate treatment group differences in change in mean number of drinks consumed from baseline to post-treatment, as indicated by the Time by Treatment Condition interaction effect
Statistical Analysis 2: Comparison: Unified Protocol vs Take Control; Test type: Superiority; p < .001, ANOVA — The threshold for significance is p <.05; Partial eta squared = .342 — This is the partial eta squared for the main effect of time
Statistical Analysis 3: Comparison: Unified Protocol vs Take Control; Test type: Superiority; p = .309, ANOVA; Partial eta squared = .018 — This is the partial eta squared for the main effect of treatment condition
Statistical Analysis 4: Comparison: Unified Protocol; After conducting the initial two-way mixed ANOVA, follow-up testing was conducted to determine the simple main effects of time (pre to post) on mean number of drinks per week within each treatment condition, which was examined using one-way repeated measures ANOVAs; Test type: Other; p < .001, ANOVA — The threshold for significance is p <.05; F = 38.92
Statistical Analysis 5: Comparison: Take Control; [analysis description as in outcome 1, analysis 4]; Test type: Other; p = .030, ANOVA; F = 5.43
Statistical Analysis 6: Comparison: Unified Protocol vs Take Control; After conducting the initial two-way mixed ANOVA, the simple main effects for treatment condition on mean number of drinks consumed per week at each timepoint (pre and post) were examined using one-way ANOVAs; Test type: Other; p = .016, ANOVA; F = 1.15 — This is the simple main effect of treatment condition on mean number of drinks consumed per week at baseline. For the UP, n=51; for the TC, n=24
Statistical Analysis 7: Comparison: Unified Protocol vs Take Control; [analysis description as in outcome 1, analysis 6]; Test type: Other; p = .007, ANOVA; F = 7.78 — This is the simple main effect of treatment condition on mean number of drinks consumed per week at post-treatment. For the UP, n=38; for the TC, n=21

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout treatment (12 or 16 sessions), up to 21 weeks, through to the 6-month follow-up.
Description: Serious adverse events were those that required immediate reporting to Boston University's Institutional Review Board according to their definitions of serious adverse events (SAEs). Percentages reflect the percent of participants who endorsed a given adverse event at any time during the trial.
Arm/Group | Unified Protocol | Take Control
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/24
Other Adverse Events (participants affected / at risk) | 0/51 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-04-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT03230006/Prot_SAP_ICF_001.pdf